CLINICAL TRIAL: NCT02903511
Title: Feasibility Study of Metformin Therapy in Autosomal Dominant Polycystic Kidney Disease.
Brief Title: Feasibility Study of Metformin Therapy in ADPKD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16-0802; R21DK107969-01A1 (NIH)
Record Dates: First submitted 2016-09-13; First posted 2016-09-16 (Estimated); Results first posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Polycystic Kidney, Autosomal Dominant
Keywords: Metformin; total kidney volume; glomerular filtration rate
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metformin (Experimental): Participants will receive metformin 500 mg tablets, starting with 1 tab twice a day. The dose will be increased by 500 mg every 2 weeks up to 1000 mg by mouth twice a day, as tolerated, for 12 months.
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator): Participants will receive placebo 500 mg tablets, starting with 1 tab twice a day. The dose will be increased by 500 mg every 2 weeks up to 1000 mg by mouth twice a day, as tolerated, for 12 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — Monitoring of safety and tolerability
  Other Names: Glucophage; Fortamet; Glumetza
  Arms: Metformin
Drug: Placebo — Monitoring of safety and tolerability
  Arms: Placebo

SUMMARY:
This study is being done to determine if treatment with metformin, a drug widely used for the treatment of diabetes type 2, is safe and well tolerated by individuals with Autosomal Dominant Polycystic Kidney Disease (ADPKD) who are not diabetic and who have slightly decreased kidney function. The study will also evaluate the effects of metformin on kidney growth and kidney function.

DETAILED DESCRIPTION:
Patients with ADPKD are still in need for a well-tolerated treatment that can be used long-term to prevent cyst growth and kidney function decline. Metformin has a long track record of a low risk-to-benefit profile in patients with diabetes or at risk for diabetes. Metformin inhibits two key processes responsible for the growth of polycystic kidneys, i.e. fluid secretion and cell proliferation, as shown in cell cultures and animal models of ADPKD. Experiments in animal models of chronic kidney disease demonstrate that metformin administration prevents kidney fibrosis and preserves kidney function. Diabetic patients who are treated with metformin appear to develop less kidney failure and live longer than patients who are treated with other anti-diabetic medications. Therefore this drug is promising for people with ADPKD, with the potential to slow cyst enlargement and preserve kidney function.

ELIGIBILITY:
Inclusion Criteria:

* Autosomal Dominant Polycystic Kidney Disease and
* An estimated glomerular filtration (GFR) rate of 50-80 ml/min/1.73 m2;
* Subject is able to sign an Informed Consent

Exclusion Criteria:

* Diabetes mellitus,
* Active infection,
* Congestive heart failure,
* Liver disease,
* Alcohol or substance dependence,
* Cigarette smoking within the last 12 months;
* Females who are pregnant or breast feeding, or
* Are unwilling to use contraception;
* Are unable to undergo magnetic resonance imaging, or
* Have a contraindication to the use of metformin

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2016-11; Primary Completion 2020-08-17 (Actual); Study Completion 2020-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Godela M Brosnahan, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Takiar V, Nishio S, Seo-Mayer P, King JD Jr, Li H, Zhang L, Karihaloo A, Hallows KR, Somlo S, Caplan MJ. Activating AMP-activated protein kinase (AMPK) slows renal cystogenesis. Proc Natl Acad Sci U S A. 2011 Feb 8;108(6):2462-7. doi: 10.1073/pnas.1011498108. Epub 2011 Jan 24. PMID 21262823
- [Background] Satriano J, Sharma K, Blantz RC, Deng A. Induction of AMPK activity corrects early pathophysiological alterations in the subtotal nephrectomy model of chronic kidney disease. Am J Physiol Renal Physiol. 2013 Sep 1;305(5):F727-33. doi: 10.1152/ajprenal.00293.2013. Epub 2013 Jul 3. PMID 23825068
- [Background] Hung AM, Roumie CL, Greevy RA, Liu X, Grijalva CG, Murff HJ, Griffin MR. Kidney function decline in metformin versus sulfonylurea initiators: assessment of time-dependent contribution of weight, blood pressure, and glycemic control. Pharmacoepidemiol Drug Saf. 2013 Jun;22(6):623-31. doi: 10.1002/pds.3432. PMID 23592561
- [Derived] St Pierre K, Cashmore BA, Bolignano D, Zoccali C, Ruospo M, Craig JC, Strippoli GF, Mallett AJ, Green SC, Tunnicliffe DJ. Interventions for preventing the progression of autosomal dominant polycystic kidney disease. Cochrane Database Syst Rev. 2024 Oct 2;10(10):CD010294. doi: 10.1002/14651858.CD010294.pub3. PMID 39356039
- [Derived] El-Damanawi R, Stanley IK, Staatz C, Pascoe EM, Craig JC, Johnson DW, Mallett AJ, Hawley CM, Milanzi E, Hiemstra TF, Viecelli AK. Metformin for preventing the progression of chronic kidney disease. Cochrane Database Syst Rev. 2024 Jun 4;6(6):CD013414. doi: 10.1002/14651858.CD013414.pub2. PMID 38837240
- [Derived] Brosnahan GM, Wang W, Gitomer B, Struemph T, George D, You Z, Nowak KL, Klawitter J, Chonchol MB. Metformin Therapy in Autosomal Dominant Polycystic Kidney Disease: A Feasibility Study. Am J Kidney Dis. 2022 Apr;79(4):518-526. doi: 10.1053/j.ajkd.2021.06.026. Epub 2021 Aug 12. PMID 34391872

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 5 participants screen failed or dropped out prior to randomization
Period: Overall Study
Arm/Group | Metformin | Placebo
Started | 26 | 25
Received Intervention | 25 | 25
Completed | 22 | 23
Not Completed | 4 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metformin | Placebo | Total
Number analyzed (Participants) | 26 | 25 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (8) | 48 (7) | 48 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 17 | 32
  Male | 11 | 8 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 26 | 24 | 50
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 26 | 25 | 51
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 26 | 25 | 51

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of Metformin
Description: Percentage of participants who at the end of 12 months are still prescribed the full randomized dose of metformin or placebo, and the percentage of participants who are prescribed at least 50% of the randomized dose
Time Frame: 12 months
Measure: Number; unit: percentage of participants
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 22 | 23
percentage of participants
  Full Dose | 50 | 100
  50% Dose | 82 | 100

2. Secondary Outcome: Change in Total Kidney Volume
Description: Total kidney volume will be measured by MRI (magnetic resonance imaging) at baseline and at 12 months. Percentage change from baseline in height-adjusted total kidney volume is reported.
Time Frame: 12 months
Population: 2 participants (1 from each group) were not analyzed due to insufficient image quality for accurate analysis.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 21 | 22
percent change | 3.45 (1.3) | 3.15 (1.61)

3. Secondary Outcome: Change in Kidney Function
Description: Estimated glomerular filtration rate (eGFR) will be calculated from serum creatinine measurements at baseline and after 3, 6, 9 and 12 months. Change from baseline at 12 months is reported.
Time Frame: 12 months
Measure: Mean (Standard Error); unit: mL/min/1.73 m^2
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 22 | 23
mL/min/1.73 m^2 | -0.41 (1.81) | -3.35 (1.70)

4. Secondary Outcome: Rate of Serious Adverse Events (SAE)
Description: Serious adverse events occurring from the time of signing informed consent until the end of the study will be monitored in both treatment arms
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 26 | 25
Participants | 2 | 0

ADVERSE EVENTS:
Time Frame: 12 Months
Arm/Group | Metformin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/25
Serious Adverse Events (participants affected / at risk) | 2/26 | 0/25
Other Adverse Events (participants affected / at risk) | 26/26 | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin (N=26) | Placebo (N=25)
Infection (Infections and infestations) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin (N=26) | Placebo (N=25)
diarrhea (Gastrointestinal disorders) | 16 (16) | 7 (7)
Nausea (Gastrointestinal disorders) | 11 (11) | 4 (4)
Vomiting (Gastrointestinal disorders) | 7 (7) | 3 (3)
Acid Reflux (Gastrointestinal disorders) | 2 (2) | 4 (4)
Light-headedness (General disorders) | 6 (6) | 4 (4)
Weakness (General disorders) | 5 (5) | 0 (0)
Viral Illness (Infections and infestations) | 5 (5) | 7 (7)
sinus infection (Infections and infestations) | 5 (5) | 2 (2)
Flatulence (Gastrointestinal disorders) | 4 (4) | 0 (0)
Abdominal cramping/pain (Gastrointestinal disorders) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-02-20): https://cdn.clinicaltrials.gov/large-docs/11/NCT02903511/Prot_SAP_000.pdf
  • Informed Consent Form (2018-05-08): https://cdn.clinicaltrials.gov/large-docs/11/NCT02903511/ICF_001.pdf